CLINICAL TRIAL: NCT00218530
Title: Naltrexone and Lofexidine in Detoxified Heroin Addicts
Brief Title: Effectiveness of Naltrexone and Lofexidine in Treating Detoxified Heroin Addicts - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-18197-1; P50-18197-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence | interventions — lofexidine

INTERVENTIONS:
Drug: Lofexidine

SUMMARY:
Stress is one of the more common reasons cited by addicts for continual drug use and relapse. Treatment approaches that target both drug-induced and stress-induced relapse may prove to be more beneficial than targeting drug-induced relapse alone. Lofexidine is a drug that reduces the physical symptoms of opiate withdrawal and may prove to have stress-reducing capabilites in drug addicts. The purpose of this study is to determine the maximal safe dose of lofexidine tolerated in naltrexone-treated heroin addicts and to find an optimal lofexidine induction schedule.

DETAILED DESCRIPTION:
Stress is one of the more common reasons cited by addicts for continual drug use and relapse. Naltrexone treatment of opiate addicts suffers from high rates of drop-out and relapse. This may be a result of naltrexone's inability to reduce symptoms of stress during early recovery. Treatment approaches that target both drug-induced and stress-induced relapse may prove to be more beneficial than targeting drug-induced relapse alone. Lofexidine is a drug that reduces the physical symptoms of opiate withdrawal and may prove to have stress-reducing capabilities. The purpose of this study is to determine the maximal safe dose of lofexidine tolerated in naltrexone-treated opiate addicts and to find an optimal lofexidine induction schedule. The study will also assess any side effects that occur during a discontinuation phase of lofexidine.

This pilot study will last a total of 8 weeks. Recently detoxified opiate dependent participants who are eligible for naltrexone treatment will enter a 4-week single-blind dose tolerability phase, during which participants will receive naltrexone and 1 of 3 twice-daily lofexidine induction schedules. All participants will be required to remain in the clinic for 2 hours immediately following dosing in order to monitor vital signs and side effects. Study visits will occur three times each week, at which time naltrexone medication for self-administration will be handed out and participants will be evaluated in terms of tolerability to treatment. After the 4 weeks of treatment, a double-blind lofexidine detoxification phase using a 5-day taper will occur. Participants will be randomly assigned to one of two maintenance-taper schedules. The first group will undergo a 5-day tapering, followed by a placebo for three weeks, followed by a 5-day tapering during Week 4. Withdrawal symptoms and side effects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for opiate dependence
* Use of heroin at least 3 times per week during the 3 months prior to entering opiate detoxification
* Documented positive urine toxicology test for opiates
* Successful initiation on naltrexone treatment as indicated by stabilization on 50 mg of naltrexone once a day
* Reads English

Exclusion Criteria:

* Regular use of anticonvulsants, sedatives/hypnotics, prescription analgesics, antihypertensives (including clonidine), antirythmics, antiretroviral medications, and tricyclic antidepressants
* Psychotic or otherwise severely psychiatrically disabled (e.g., suidical, homicidal, currently manic)
* Abstinent from opiates for more than four weeks prior to naltrexone initiation
* Any medical problems that might make naltrexone treatment unsafe, such as hepato-cellular injury as evidenced by abnormal liver enzyme tests (including SGOT, SGPT, and GGT levels greater than three times normal) and a history of cirrhosis
* Hypotension with a resting blood pressure below 90/50 mm Hg
* Pregnant, breastfeeding, or refusal to use a reliable form of contraception throughout the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 2003-03; Study Completion 2004-09

PRIMARY OUTCOMES:
Retention in treatment; measured throughout 8 weeks
Frequency and amount of opiate use; measured weekly
Stress levels; measured weekly

SECONDARY OUTCOMES:
Tolerability; measured throughout 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, M.D., Principal Investigator — Yale University
Locations (1):
- Substance Abuse Treatment Unit, New Haven, Connecticut, United States